CLINICAL TRIAL: NCT03980626
Title: Study on Physical Activity's Relationship With Cancer and Cognition: A Pilot Randomized Trial
Brief Title: Study on Physical Activity's Relationship With Cancer and Cognition
Acronym: SPARCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0091-19-FB
Record Dates: First submitted 2019-05-28; First posted 2019-06-10 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Breast Neoplasm Female
Keywords: physical activity; exercise; cognition; brain health; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Intervention (Experimental): Walking participants will engage in the 3-times weekly walking program for 12 weeks.
  Interventions: Behavioral: Walking
- Usual Care (No Intervention): Usual care participants will be offered two personalized exercise sessions with a trained exercise specialist after all post-intervention data have been collected.

INTERVENTIONS:
Behavioral: Walking — The exercise intervention is designed to improve cardiorespiratory fitness, a known correlate of cognition and brain health, and follows the American College of Sports Medicine exercise guidelines for cancer survivors. Participants will engage in small group, moderate-to-vigorous intensity walking sessions three times weekly. Sessions will begin with a warm-up and end with a cool down and be progressive in nature. Volume of exercise will increase across weeks such that participants will progress from 15-20 minutes of walking to 40-45 minutes by week 8, and from 40-55% of their estimated heart rate reserve (HRR) to 65% of their HRR by week 9. All sessions will be led by trained exercise specialists to ensure close monitoring of participant safety. Participants will wear heart rate monitors and be asked to rate their perceived exertion to ensure they are exercising within the prescribed range. Modifications to each participant's exercise prescription will be made as needed.
  Other Names: Aerobic Exercise Training
  Arms: Walking Intervention

SUMMARY:
This pilot study tests the effects of aerobic exercise training on cognitive function in breast cancer survivors (BCS). Participants will be randomized to a 12-week walking intervention or usual care. Walking participants will attend small group sessions led by an exercise specialist 3 times weekly. Usual care participants will complete baseline and post-testing and be offered two sessions with an exercise specialist. All participants will complete a fitness test, electrophysiology, and patient-reported outcomes at baseline and post-intervention. A subset of participants will also be invited to undergo magnetic resonance imaging (MRI). The investigators will generate preliminary data on clinical and biological correlates of exercise and cognition, including treatment protocol, cardiorespiratory fitness, brain structure and function, and cancer-related fatigue.

DETAILED DESCRIPTION:
Aim 1: This pilot study tests the effects of aerobic exercise training on cognitive function in breast cancer survivors (BCS). To test aim 1, the investigators will randomize up to forty post-menopausal BCS (3-24 months post-treatment) to a 12-week walking intervention (n=20) or usual care (n=20). Walking participants will attend small group (n=3-5 BCS) sessions led by an exercise specialist 3 times weekly. Usual care participants will complete baseline and post-testing and be offered two sessions with an exercise specialist after all data have been collected. Aim 1 measures include accelerometry, neurocognitive testing, and patient-reported outcomes at baseline and post-intervention.

Aim 2: The investigators will generate preliminary data on clinical and biological correlates of exercise and cognition, including treatment protocol, cardiorespiratory fitness, brain structure and function, and cancer-related fatigue. To test aim 2, all participants will complete a fitness test, electrophysiology, and patient-reported outcomes at baseline and post-intervention. A subset of participants will also be invited to undergo magnetic resonance imaging (MRI).

Data will be analyzed using descriptive statistics and analysis of covariance, and effect sizes expressed as standard mean difference will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Post-menopausal at time of diagnosis
* First, primary diagnosis of Stage I-IIIa breast cancer
* Completed treatment 3-24 months prior to study start
* Available to attend exercise sessions 3 times weekly for 12 weeks
* No scheduled travel >7 consecutive days during the intervention
* Agree to be randomized
* Willingness to wear, charge, and sync Fitbit
* English reading and speaking
* Physician's clearance to exercise
* Provide written informed consent

Exclusion Criteria:

* Males
* Pre- or peri-menopausal at the time of diagnosis
* Stage 0 or metastatic disease
* Currently receiving chemotherapy or radiation therapy
* More than 24 months post-treatment
* Scheduled to receive breast surgery
* Second cancer diagnosis (excluding non-invasive skin cancers)
* Self-report an average of ≥60 minutes of moderate to vigorous physical activities (MVPA) per week for the previous 6 months
* Not cleared to exercise by a physician
* Not available to attend 3 times weekly exercise sessions for 12 weeks
* Out of town travel scheduled for >1 week during the intervention
* Unwilling to complete baseline assessments
* Unwilling to be randomized to the exercise or control group
* Unwilling to wear, charge, and sync the Fitbit during the study period
* Unable to read and speak in English
* Unwilling to provide written informed consent to participate
* Cognitive impairment prior to baseline assessment
* History of stroke, transient ischemic attack, other neurological disorders, or brain surgery involving tissue removal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Executive Function | Baseline, Week 12
  A comprehensive neurocognitive battery will be administered to measure executive function as defined by a latent factor of manifest indicators of performance on executive function tasks.
Change in Working Memory | Baseline, Week 12
  A comprehensive neurocognitive battery will be administered to measure working memory as defined by a latent factor of manifest indicators of performance on working memory tasks.
Change in Processing Speed | Baseline, Week 12
  A comprehensive neurocognitive battery will be administered to measure processing speed as defined by a latent factor of manifest indicators of processing speed tasks.

SECONDARY OUTCOMES:
Regional brain volume | Baseline, Week 12
  Magnetic Resonance Imaging (MRI) will be used to measure regional volume.
White matter structural integrity | Baseline, Week 12
  Diffusion tensor imaging (DTI) will be used to measure white matter structural integrity (fractional anisotropy, diffusivity).
Resting state functional connectivity | Baseline, Week 12
  Resting state function MRI will be used to measure resting state functional connectivity (patterns of blood oxygen level dependent (BOLD) activity within seed regions of interest compared to whole brain activity).
N2pc Amplitude | Baseline, Week 12
  N2pc amplitude is a neural measure of spacial attention during the Visual Search Task (measured in microvolts) to be measured with electroencephalography (Visual Search Task, Change Detections Task).
Cardiorespiratory Fitness | Baseline, Week 12
  Fitness will be measured with a submaximal exercise test. The Naughton Protocol for submaximal graded exercise tests will be used to examine change in cardiovascular fitness.
Cancer-related Fatigue | Baseline, Week 12
  The Functional Assessment in Chronic Illness Therapy (FACIT) - Fatigue Scale will be used to measure cancer-related fatigue. Scores range from 0-52, with higher scores indicating less cancer-related fatigue.
Objective Activity Behavior | Baseline, Week 12
  Objective activity behavior (average minutes per day) will be measured using actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Diane K Ehlers, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request as required by journal publishers during dissemination phase of the study.
Time Frame: When summary data are published.
Access Criteria: Individual participant data (IPD) will be provided as required by journals in which summary data are published.

REFERENCES:
- [Derived] Page LL, Fanning J, Phipps C, Berger A, Reed E, Ehlers D. Heart Rate Monitoring Among Breast Cancer Survivors: Quantitative Study of Device Agreement in a Community-Based Exercise Program. JMIR Cancer. 2024 Jun 20;10:e51210. doi: 10.2196/51210. PMID 38900505